CLINICAL TRIAL: NCT04907110
Title: The Effects of Exercise Training Combined With NR Supplementation on Metabolic Health in Older Individuals
Brief Title: NR Supplementation and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL77756.068.21
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Overweight and Obesity; Aging; Type 2 Diabetes
Keywords: exercise; NR supplementation; NAD metabolism
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2; Motor Activity | interventions — nicotinamide-beta-riboside; Exercise

STUDY DESIGN:
Intervention Model Description: The present study is a randomized, double-blinded, placebo-controlled double arm longitudinal intervention study in a pre and post design.
Who Masked: Participant, Investigator
Masking Description: Participants and Investigator will be blinded for the study material (i.e. NR or placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + NR (Experimental): Participants will be asked to take two pills of NR (250mg/pill) twice daily (a total of 4 pills/day; 1000mg/day), for 40 days. During days 17-38 of the NR intervention, participants will perform a 3-weeks supervised exercise training program with four ~30 min exercise sessions per week (two endurance session on a bike at 70%Wmax and two high intensity interval (HIIT) sessions. To assess the outcomes, participants will undergo three test days before the start of the NR supplementation and repeat these three test days at the end (day 38-40) of NR supplementation.
  Interventions: Dietary Supplement: Niagen; Other: Exercise
- Exercise + Placebo (Placebo Comparator): Participants will be asked to take two pills of placebo, twice daily (a total of 4 pills/day), for 40 days. During days 17-38 of the intervention, participants will perform a 3-weeks supervised exercise training program with four ~30 min exercise sessions per week (two endurance session on a bike at 70%Wmax and two high intensity interval (HIIT) sessions. To assess the outcomes, participants will undergo three test days before the start of the NR supplementation and repeat these three test days at the end (day 38-40) of the placebo supplementation.
  Interventions: Other: Exercise

INTERVENTIONS:
Dietary Supplement: Niagen — Participants in the NR supplementation + exercise group will undergo oral NR supplementation for 40 days. NiagenTM is the name for the dietary supplement containing NR (ChromaDex, Inc. Irvine, USA). The total dosage of NR per day will be 1000mg. This supplementation time of 40 days 1000mg/day
  Other Names: Nicotinamide Riboside (NR)
  Arms: Exercise + NR
Other: Exercise — During days 17-38 of the NR/placebo intake, participants will perform a 3-weeks supervised exercise training program with four ~30 min exercise sessions per week (two endurance session on a bike at 70%Wmax and two high intensity interval (HIIT) sessions.

SUMMARY:
The number of age-related chronic diseases (like obesity, type 2 diabetes and cardiovascular diseases) is increasing rapidly worldwide, reaching pandemic proportions. These age-related chronic diseases are associated with metabolic disturbances and mitochondrial dysfunction in humans. Nicotinamide adenosine dinucleotide (NAD) levels play an important role in energy metabolism and mitochondrial functioning and indeed it has been shown that high concentrations of NAD+ as well as a high NAD+/NADH ratio are strongly associated with metabolic and mitochondrial health. In contrast, decreased NAD+ bioavailability is reported in both ageing and obese humans as well as in diabetic mice. These findings fueled the idea of influencing NAD+ bioavailability in order to improve metabolic disturbances and mitochondrial dysfunction in humans. Supplementation with nicotinamide riboside (NR), a naturally occurring form of vitamin B3, may provide a way to boost cellular NAD+ levels. However, in contrast to animal studies, NR supplementation in humans has so far been unsuccessful in improving skeletal muscle mitochondrial function, exercise capacity or insulin sensitivity. Recently, it has been suggested that a situation where NAD+ levels become limited, is needed for NR supplementation to exert beneficial health effects. This situation could be achieved by combining exercise and NR supplementation. However, studies combining NR and exercise are lacking, which is why we would like to perform such a study here.

DETAILED DESCRIPTION:
Rationale: The number of age-related chronic diseases (like obesity, type 2 diabetes and cardiovascular diseases) is increasing rapidly worldwide, reaching pandemic proportions. These age-related chronic diseases are associated with metabolic disturbances and mitochondrial dysfunction in humans. Nicotinamide adenosine dinucleotide (NAD) levels play an important role in energy metabolism and mitochondrial functioning and indeed it has been shown that high concentrations of NAD+ as well as a high NAD+/NADH ratio are strongly associated with metabolic and mitochondrial health. In contrast, decreased NAD+ bioavailability is reported in both ageing and obese humans as well as in diabetic mice. These findings fueled the idea of influencing NAD+ bioavailability in order to improve metabolic disturbances and mitochondrial dysfunction in humans. Supplementation with nicotinamide riboside (NR), a naturally occurring form of vitamin B3, may provide a way to boost cellular NAD+ levels. However, in contrast to animal studies, NR supplementation in humans has so far been unsuccessful in improving skeletal muscle mitochondrial function, exercise capacity or insulin sensitivity. Recently, it has been suggested that a situation where NAD+ levels become limited, is needed for NR supplementation to exert beneficial health effects. This situation could be achieved by combining exercise and NR supplementation. However, studies combining NR and exercise are lacking, which is why we would like to perform such a study here.

Objective: The primary objective of this study is to determine whether combined treatment of exercise and NR imposes greater improvements in skeletal muscle mitochondrial metabolism in older humans compared to exercise treatment alone. The secondary objective is to determine whether combined treatment of exercise and NR supplementation imposes greater improvements in sleeping metabolic rate (SMR). As explorative objectives, we will examine whether combined treatment with exercise and NR imposes greater improvements in muscle (NAD) metabolites, energy metabolism and physical performance.

Study design: The present study is a randomized, double-blinded, placebo-controlled double arm longitudinal intervention study in a pre and post design.

Study population: 30 older male and (postmenopausal) female participants, aged 65 - 80 years with a BMI between 25-35 kg/m2 will perform this study (15 participants in the exercise+placebo group, 15 participants in the exercise+NR group). From experience with similar studies, we estimate a drop-out rate of 20% and a screening failure of 50% (due to the strict inclusion criteria), resulting in maximally 36 subjects that have to be included and 72 subjects that have to be screened (maximally).

Intervention (if applicable): Participants will be asked to take two pills of NR (250mg/pill), or placebo, twice daily (two with breakfast and two with diner, a total of 4 pills/day; 1000mg/day), for 40 days. During days 17-38 of the NR intervention, participants will perform a 3-weeks supervised exercise training program with four ~30 min exercise sessions per week (two endurance session on a bike at 70%Wmax and two high intensity interval (HIIT) sessions. Participants will be randomly assigned to the placebo + exercise or NR + exercise arm. To assess the outcomes, participants will undergo three test days before the start of the NR supplementation and repeat these three test days at the end (day 38-40) of NR supplementation.

Main study parameters/endpoints: The primary study endpoints is ex vivo skeletal muscle mitochondrial function measured via high-resolution respirometry. Explorative objectives are muscle (NAD) metabolites, energy metabolism and physical performance.

ELIGIBILITY:
Inclusion Criteria:

* Participants are able to provide signed and dated written informed consent prior to any study specific procedures
* Aged ≥ 65 and ≤ 80 years
* Body mass index (BMI) 25 - 35 kg/m2
* Stable dietary habits (no weight loss or gain > 5 kg in the past 3 months)
* No signs of active cardiovascular disease, liver or kidney malfunction

Exclusion Criteria:

* Type 2 diabetes
* Patients with congestive heart failure and and/or severe renal and or liver insufficiency
* Uncontrolled hypertension
* Any contra-indication for MRI scanning
* Alcohol consumption of >3 servings per day for man and >2 servings per day for woman
* Smoking
* Unstable body weight (weight gain or loss > 5kg in the last 3 months)
* Engagement in structured exercise activities > 2 hours a week
* Previous enrolment in a clinical study with an investigational product during the last 3 months or as judged by the Investigator which would possibly hamper our study results
* Medication use known to hamper subject's safety during the study procedures
* Subjects who do not want to be informed about unexpected medical findings
* Use of food supplements containing NR or Resveratrol (similar working mechanisms)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Ex vivo muscle mitochondrial function | Pre-intervention test day 3 + day 40 of the intervention NR/Placebo + exercise
  Ex vivo mitochondrial function in skeletal muscle measured by oxygen consumption in muscle fibres (muscle biopsy vastus lateralis) on lipid-derived and carbohydrate-derived substrates.

SECONDARY OUTCOMES:
Maximal aerobic capacity | Pre-intervention test day 1 + Day 38
  Maximal aerobic capacity measured during a VO2max cycling test in ml/kg/min
Physical performance | Pre-intervention test day 1 + Day 38
  Physical performance is measured during a 6-minute walk test (6MWT) expressed as the distance covered during 6 minutes walking as well as the time necessary to stand up from a chair (TCST).
Skeletal muscle NAD concentrations (ex-vivo) | Pre-intervention test day 3 + Day 40
  Skeletal muscle NAD metabolites are measured in muscle biopsies using metabolomics
Skeletal muscle NAD concentration (in-vivo) | Pre-intervention test day 3 + Day 40
  Skeletal muscle NAD metabolites are measured in vivo using phosphorus magnetic resonance spectroscopy in the m. vastus lateralis.
Intrahepatic lipid content | Pre-intervention test day 1 + Day 38
  Intrahepatic lipid content is measured using proton magnetic resonance spectroscopy
Upper leg muscle mass | Pre-intervention test day 1 + Day 38
  Upper leg muscle mass is measured with magnetic resonance imaging
Body composition | Pre-intervention test day 1 + Day 38
  Body composition is measured using the BodPod technique and fat mass (kg and %) and fat-free mass (kg) will be determined.
Quality of life | Pre-intervention test day 1 + Day 38
  Quality of life will be assessed by a questionnaire (in arbitrary units measured via the 32-item survey)
Blood metabolites | Pre-intervention test day 3 + Day 40
  Metabolites in the blood (i.e. glucose, free fatty acids, triglycerides, cholesterol, insulin in mmol/L taken via a venepuncture)
Submaximal exercise energy expenditure | Pre-intervention test day 3 + Day 40
  Submaximal exercise energy expenditure will be measured via indirect calorimetry during a 60-minute submaximal cycling exercise at 50% Wmax
Sleeping metabolic rate | Pre-intervention test day 2 + Day 39
  Sleeping metabolic rate will be measured during a 11 hour stay in a respiration chamber via indirect calorimetry
Exercise efficiency | Pre-intervention test day 3 + Day 40
  Exercise efficiency will be measured during a 60-minute submaximal cycling test via indirect calorimetry in kJ/min

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data can be obtained with the principal investigator if desired.